CLINICAL TRIAL: NCT00857623
Title: A Phase IIa, Double-Blind, Randomised, Parallel-Group, Multi-Centre Study to Evaluate the Analgesic Efficacy of 28 Days' Oral Administration of AZD2066 Compared With Placebo in Patients With Painful Diabetic Neuropathy
Brief Title: Study to Evaluate the Analgesic Efficacy of 28 Days' Oral Administration of AZD2066 Compared With Placebo in Patients With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0475C00009
Record Dates: First submitted 2009-02-27; First posted 2009-03-06 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Pain; Diabetic Neuropathy
Keywords: Pain; Diabetic Neuropathy; PDN; Analgesia; Efficacy
MeSH Terms: conditions — Pain; Diabetic Neuropathies; Agnosia | interventions — AZD2066

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD2066
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2066 — Capsule, once daily, 12 mg AZD2066 day 1-4 and 18 mg AZD2066 day 5-28.
  Arms: 1
Drug: Placebo — Capsule, once daily
  Arms: 2

SUMMARY:
The purpose of this study is to investigate if AZD2066 can relieve the pain arising from painful diabetic neuropathy compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Clinical diagnosis of painful diabetic neuropathy.
* non-fertile females

Exclusion Criteria:

* Other pain that may confound assessment of neuropathic pain.
* Ongoing significant peripheral arterial diseases, skin ulcers, or amputation in the lower extremities.
* History of psychotic disorders among first degree relatives.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Lilja, Study Director — AstraZeneca R&D Södertälje151 85 Södertälje, Sweden; Charles E Argoff, MD, Principal Investigator — Albany Medical , NY 12208, USA
Locations (19):
- United States (19):
  - Reserach Site, Bella Vista, Arkansas
  - Research Site, National City, California
  - Research Site, Walnut Creek, California
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Madisonville, Kentucky
  - Research Site, Owing Mills, Maryland
  - Research Site, Bingham Farms, Michigan
  - Research Site, Willingboro, New Jersey
  - Reasearch Site, Albany, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Indiana, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted between February 2009 and August 2009in the United States.
Pre-assignment Details: The study consisted of a 42-day enrollment phase (including washout and baseline period), a 28-day treatment phase (10-day inpatient and 18-day outpatient) where patients were randomized to AZD2066 or placebo, and a 7-day follow-up phase. Patients randomized to treatment with AZD2066 received 12 mg from Days 1 to 4 and 18 mg from Days 5 to 28.
Groups:
- AZD2066: Capsule, once daily. 12 mg AZD2066 day 1-4 and 18 mg AZD2066 day 5-28.
Period: Overall Study
Arm/Group | AZD2066 | Placebo
Started | 62 | 65
Completed | 48 | 55
Not Completed | 14 | 10
Not completed — Adverse Event | 5 | 2
Not completed — Study-specific discontinuation criteria | 5 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Severe non-compliance to protocol | 1 | 1
Not completed — Intake of prohibited medication | 0 | 1
Not completed — Positive for HEP C | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- AZD2066: Capsule, once daily 12 mg AZD2066 day 1-4 and 18 mg AZD2066 day 5-28
- Total: Total of all reporting groups
Arm/Group | AZD2066 | Placebo | Total
Number analyzed (Participants) | 62 | 65 | 127
Age Continuous [Mean (Standard Deviation); unit: years] — All randomized patients.
  years | 59.2 (9.2) | 57.0 (8.7) | 58.1 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants] — All randomized patients.
  Participants
    Female | 26 | 31 | 57
    Male | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Numerical Rating Scale (NRS) Score From Baseline to Last 5 Days of Treatment
Description: Change of mean pain intensity from 5-day baseline to the last 5 days of treatment, measured twice daily with NRS (12 hours recall).
  Mean pain intensity for 5-day baseline period (evening Day -6 to moning Day-1) and mean pain intensity for last 5 days on treatment (ie, last dose day and the 4 preceding calendar days) was calculated based on the numerical rating scale (NRS)(0-10). 0=No pain, 10=Worst pain imaginable.
Time Frame: From baseline to day 28
Population: Per Protocol population (PP)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Scores on a scale | -2.33 (0.37) | -2.52 (0.36)

2. Secondary Outcome: Daily Numerical Rating Scale (NRS) Pain Scores and Change From Baseline Over Time to Day 28.
Description: Mean pain intensity per day (mean of morning and evening NRS values) and change from baseline were calculated for each study day. Baseline value= mean pain intensity for the 5-day baseline period. NRS scale (0- 10) where 0= No pain and 10= Worst pain imaginable.
Time Frame: From baseline to 28 days
Population: Per Protocol population (PP)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Scores on a scale | -2.3 (2.2) | -2.5 (2.3)

3. Secondary Outcome: Number of Patients With >=30% Reduction From Baseline in Numerical Rating Scale (NRS) Pain Intensity Score at Day 28
Description: Pain intensity score reduction=(change from baseline at D28/baseline)*100 Responder= pain intensity score reduction ≥30% (yes/no)? Responder rate= (no. of responders/total no. of patients)*100
Time Frame: 28 days
Population: Per Protocol population (PP)
Measure: Number; unit: Participants
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Participants | 23 | 25

4. Secondary Outcome: Number of Patients With >=50% Reduction From Baseline in Numerical Rating Scale (NRS) Pain Intensity Score at Day 28
Description: Pain intensity score reduction= (change from baseline D28/baseline)*100 Responder=pain intensity score reduction ≥50% (Yes/No)? Responder rate= (no. of responders/total no. of patients)*100
Time Frame: 28 days
Population: Per Protocol population (PP)
Measure: Number; unit: Participants
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Participants | 15 | 15

5. Secondary Outcome: Number of Patients With Patient Global Impression of Change (PGIC) Score of at Least "Much Improved" at Day 28.
Description: Patient Global Impression of Change (PGIC) scale ranges from 1-7, where 1= Very much improved and 7= Very much worse.
  Responder= Patient with a response of "much improved" or "very much improved" Responder rate= (no. of responders/total no. of patients)*100
Time Frame: 28 days
Population: Per Protocol population (PP)
Measure: Number; unit: Participants
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Participants | 20 | 28

6. Secondary Outcome: Change in McGill Pain Questionnaire Short Form (MPQ-SF) Sensory Index From Baseline to Day 28.
Description: Sensory index= sum of the intensity scale values of the words chosen for the descriptors 1-11 in the questionnaire. Range of scores for the sensory index= 0-33 (higher score represents a worse condition).
  Change from baseline (measured prior to randomization) to Day 28 was calculated.
Time Frame: From baseline to day 28.
Population: Per Protocol population (PP)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Scores on a scale | -6.87 (0.93) | -7.68 (0.88)

7. Secondary Outcome: Change in McGill Pain Questionnaire Short Form (MPQ-SF) Affective Index From Baseline to Day 28.
Description: Affective index= sum of the intensity scale values of the words chosen for the descriptors 12-15 in the questionnaire. Range of scores for the affective index=0-12 (higher score represents a worse condition).
  Change from baseline (measured prior to randomization) to Day 28 was calculated.
Time Frame: From baseline to day 28.
Population: Per Protocol population (PP)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Scores on a scale | -1.87 (0.35) | -2.06 (0.34)

8. Secondary Outcome: Change in Brief Pain Inventory-Short Form (BPI-SF) Pain Severity From Baseline to Day 28.
Description: Change from baseline (measured prior to randomization) to Day 28 was calculated for the pain severity (mean of 4 intensity items). Each intensity item is recorded on a Numerical rating Scale (NRS) 0-10, where 0=No pain and 10= The worst pain.
Time Frame: From baseline to day 28..
Population: Per Protocol population (PP)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Scores on a scale | -1.99 (0.35) | -2.19 (0.34)

9. Secondary Outcome: Change in Brief Pain Inventory-Short Form (BPI-SF) Pain Interference From Baseline to Day 28.
Description: Change from baseline (measured prior to randomization) to Day 28 was calculated for pain interference (mean of 7 interference items). Each interference item is recorded on a Numerical Rating Scale (NRS 0-10), where 0= No interference and 10= Interferes completely.
Time Frame: From baseline to 28 days
Population: Per Protocol population (PP)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | AZD2066 | Placebo
Number analyzed (Participants) | 46 | 51
Scores on a scale | -2.13 (0.31) | -2.13 (0.30)

ADVERSE EVENTS:
Arm/Group | AZD2066 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/62 | 1/65
Other Adverse Events (participants affected / at risk) | 19/62 | 20/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2066 (N=62) | Placebo (N=65)
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Cardiac failure congestive; Myocardial infarction (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2066 (N=62) | Placebo (N=65)
Headache (Nervous system disorders) | 9 | 11
Dizziness (Nervous system disorders) | 7 | 4
Diarrhea (Gastrointestinal disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other